CLINICAL TRIAL: NCT00528619
Title: Phase I Study Of SU011248 In Combination With Pemetrexed, Pemetrexed/Cisplatin And Pemetrexed/Carboplatin In Patients With Advanced Solid Malignancies
Brief Title: A Study To Find The Best Dose Of SU011248 When Given With Pemetrexed, Pemetrexed And Cisplatin Or Pemetrexed And Carboplatin In Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6181084
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-04

CONDITIONS: Neoplasms
Keywords: Solid tumor malignancy; non-small cell lung cancer; sunitinib; pemetrexed; Phase 1; Mesothelioma
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Mesothelioma | interventions — Sunitinib; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Sunitinib, Pemetrexed, Cisplatin, Carboplatin

INTERVENTIONS:
Drug: Sunitinib, Pemetrexed, Cisplatin, Carboplatin — Dose finding study using Sunitinib daily by oral capsule in a continuous regimen or administered for 2 weeks out of every 3 weeks, with pemetrexed every 3 weeks or also with cisplatin 75 mg/m2 or carboplatin AUC=5 mg*min/mL until progression or unacceptable toxicity.
  Other Names: Sutent, SU011248, Alimta, Platinol, Paraplatin

SUMMARY:
This study will assess the maximum tolerated dose, overall safety and antitumor activity of SU011248 in combination with pemetrexed, pemetrexed and cisplatin or pemetrexed and carboplatin in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of a solid cancer which is not responsive to standard therapy or for which no standard therapy exists.
* Patient has a good performance status (ECOG 0 or 1).

Exclusion Criteria:

* Prior treatment with either pemetrexed or SU011248.
* Coughing up blood within 4 weeks before starting study treatment (small amounts okay).
* Hypertension that cannot be controlled by medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2006-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To determine maximally tolerated dose of SU011248 (dosed continuously or on a 2/1 Schedule) when given in combination with pemetrexed, pemetrexed and cisplatin or pemetrexed and carboplatin. | From screening until at least 28 days beyond discontinuation of study treatment

SECONDARY OUTCOMES:
To evaluate the plasma pharmacokinetics of SU011248 and its metabolite, SU012662 in addition to pemetrexed, SU011248 and pemetrexed/cisplatin, and SU011248 and pemetrexed/carboplatin when these drugs are co-administered. | From screening until disease progression or discontinuation of the study
To preliminarily assess the antitumor activity of SU011248 in addition to pemetrexed, SU011248 and pemetrexed/cisplatin, and SU011248 and pemetrexed/carboplatin in patients with non-small cell lung cancer or advanced unresectable mesothelioma. | From screening until disease progression or discontinuation of the study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Pfizer Investigational Site, Aurora, Colorado, United States
- Canada (2):
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Montreal, Quebec